CLINICAL TRIAL: NCT00359918
Title: Randomized, Controlled Multicenter Trial of Prehospital Initiated Facilitated PCI Versus Primary PCI in Patients With STEMI LIPSIA-STEMI Trial
Brief Title: Randomized Multicenter Trial of Prehospital Initiated Facilitated Percutaneous Coronary Intervention (PCI) Versus Primary PCI in ST-segment-Elevation MI (STEMI)
Acronym: LIPSIA STEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Holger Thiele (Other)
Responsible Party: Sponsor-Investigator, Holger Thiele, PI, University of Leipzig
Organization: University of Leipzig (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reg.-Nr. 008/2006
Record Dates: First submitted 2006-08-01; First posted 2006-08-03 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Myocardial Infarction
Keywords: infarction; facilitated PCI; primary PCI; infarct size; fibrinolysis; ST-elevation myocardial infarction (STEMI)
MeSH Terms: conditions — Myocardial Infarction; Infarction; ST Elevation Myocardial Infarction | interventions — Fibrinolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prehospital facilitated PCI (Experimental)
  Interventions: Drug: fibrinolysis
- Primary PCI (Active Comparator)
  Interventions: Procedure: Primary PCI

INTERVENTIONS:
Drug: fibrinolysis — Primary PCI
  Other Names: Primary PCI
  Arms: Prehospital facilitated PCI
Procedure: Primary PCI — Primary PCI
  Arms: Primary PCI

SUMMARY:
Prehospital initiated facilitation of primary percutaneous coronary intervention by fibrinolysis might be helpful in re-opening the infarct related artery prior to percutaneous coronary intervention.

This studies tests the hypothesis that prehospital initiated facilitated PCI is superior to primary percutaneous coronary intervention with respect to infarct size.

DETAILED DESCRIPTION:
Patients with STEMI with symptoms < 3 hours are randomized in the region of Leipzig to either prehospital full-dose fibrinolysis (+ASA, Clopidogrel and heparin) with subsequent facilitated percutaneous coronary intervention or to primary percutaneous coronary intervention (after ASA + heparin + clopidogrel).

Patients undergo cardiac magnetic resonance for assessment of infarct size early at day 1-4 after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Angina pectoris < 3 hours
* ST-elevation myocardial infarction

Exclusion Criteria:

* Active bleeding
* Active gastric ulcus
* Previous stroke
* Uncontrolled hypertension (> 200 mmHg)
* Cerebral surgery < 8 weeks
* Major surgery < 4 weeks
* Malignancy
* Treatment with coumarines
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Infarct size and microvascular obstruction assessed by MRI | 1-6 days

SECONDARY OUTCOMES:
Clinical endpoints (bleeding, death, Re-MI, stroke) | 30 days
ST-segment resolution | 90 min

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, PhD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] de Waha S, Eitel I, Desch S, Fuernau G, Lurz P, Stiermaier T, Blazek S, Schuler G, Thiele H. Prognosis after ST-elevation myocardial infarction: a study on cardiac magnetic resonance imaging versus clinical routine. Trials. 2014 Jun 25;15:249. doi: 10.1186/1745-6215-15-249. PMID 24962156
- [Derived] Thiele H, Eitel I, Meinberg C, Desch S, Leuschner A, Pfeiffer D, Hartmann A, Lotze U, Strauss W, Schuler G; LIPSIA-STEMI Trial Group. Randomized comparison of pre-hospital-initiated facilitated percutaneous coronary intervention versus primary percutaneous coronary intervention in acute myocardial infarction very early after symptom onset: the LIPSIA-STEMI trial (Leipzig immediate prehospital facilitated angioplasty in ST-segment myocardial infarction). JACC Cardiovasc Interv. 2011 Jun;4(6):605-14. doi: 10.1016/j.jcin.2011.01.013. PMID 21700245